CLINICAL TRIAL: NCT05656937
Title: Oblique Versus Transverse Transducer Orientation Approach for Ultrasound Guided Internal Jugular Venous Cannulation in Heart Surgery Pediatric Patients
Brief Title: Oblique Versus Transverse Orientation Approach for Internal Jugular Venous Cannulation in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aldy Heriwardito, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IndonesiaUAnes109
Record Dates: First submitted 2021-07-18; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Heart; Surgery, Heart, Functional Disturbance as Result; Pediatric ALL
Keywords: oblique orientation; transverse orientation; internal jugular venous cannulation; ultrasound guided; short axis; oblique axis
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oblique orientation (Experimental): cannulation will be oblique approach
  Interventions: Procedure: internal jugular venous cannulation
- transverse approach (Active Comparator): cannulation will be transverse approach
  Interventions: Procedure: internal jugular venous cannulation

INTERVENTIONS:
Procedure: internal jugular venous cannulation — internal jugular venous cannulation

SUMMARY:
this study aimed to compare oblique versus transverse orientation approach in jugular venous cannulation in term of cannulation success in pediatric heart surgery patients

DETAILED DESCRIPTION:
Sixty patients randomised into two groups, 30 patients in experimental group (oblique orientation) and 30 patients in control group (transverse orientation). All cannulation took place in the operation room. Patients underwent general anesthesia and placed in supine position. Standard monitoring (electrocardiogram, non-invasive arterial pressure, pulseoxymetry) was carried out during the procedure for all patients. Before preparation of the skin, a pre-procedure ultrasound examination was performed to verify internal jugular vein patency, and its diameter was measured. Once the side had been chosen, the cannulation was performed following a sterile technique. All procedure were performed by Seldinger technique, with 22 Gauge IV catheter attached with 3 ml syringe as introducer needle. The vascular puncture was performed under ultrasound guidance, using a single-person technique. With transverse orientation, the transducer was placed transversally over the neck, and once the vein was visible in the middle of the ultrasound image, the needle was inserted in the plane perpendicular to the long axis of the transducer. With oblique orientation, the operator first obtained a transverse view of the vein and then rotated the transducer to 45 degrees (midway) between transverse and longitudinal view.

ELIGIBILITY:
Inclusion Criteria:

* patients age 3 months to 12 years old, weight 5-20 kg, male or female
* who undergo heart surgery and indicated to have central venous cannulation
* American Society of Anesthesiologist Physical Class 1-3
* Family or representation of the patients agreed to participate in this study and sign informed consent

Exclusion Criteria:

* history of surgery in the area of cannulation
* already placed central venous cannulation <72 hours in the same venous
* sign of infection, hematoma, emphysema, in the area of cannulation
* history of cervical trauma
* severe hemostatic disorder (International Normalized Ratio>2, thrombocyte <50.000, Prothrombin time>1.5 times, Activated Partial Thromboplastin Time > 1.5 times

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
% of patients with successful cannulation in first attempt | at the procedure of cannulation
  The number of patients undergo cannulation with first attempt success are shown in percentage

SECONDARY OUTCOMES:
% of patients with successful cannulation with designed approach | at the procedure of cannulation
  The number of patients undergo cannulation using designed approach are shown in percentage

CONTACTS AND LOCATIONS:
Overall Officials: aldy heriwardito, Doctor, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided